CLINICAL TRIAL: NCT06127784
Title: Survivorship After Head and Neck Cancer: A Randomized Controlled Trial Evaluating Patient Care and Adherence to Follow-up
Brief Title: Survivorship After HNC: A Randomized Controlled Trial Evaluating Patient Care and Adherence to Follow-up
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Danielle MacNeil, Doctor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 123657
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Head and Neck Cancer; Survivorship
Keywords: Motivational Interviewing; Counselling; Survivorship Care Plan; Treatment Adherence
MeSH Terms: conditions — Head and Neck Neoplasms; Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: A prospective, randomized controlled trial at a single centre with 2 groups of 88 adults. The intervention group will receive a one-hour treatment summary and survivorship care plan (TSSP) intervention specifically tailored to the needs of head and neck cancer patients delivered within a motivational interviewing counselling session with a clinical nurse specialist. The standard care group will receive standard of care treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MI Counselling (Experimental): An individualized treatment summary and survivorship care plan (TSSP) will be prepared within a one-hour motivational interviewing (MI) counseling session with a clinical nurse specialist. Participants will be asked to identify their top three symptom/survivorship concerns. The intervention will address symptoms/survivorship care specifically tailored to the needs of head and neck cancer patients based on the best available evidence and consultation with patients and a multidisciplinary team of head and neck cancer specialists. Patient participants will engage in role play to empower them to follow-up with their healthcare provider regarding their survivorship care needs.
  Interventions: Other: Motivational interviewing counselling session
- Standard care (No Intervention): The standard care group will receive no intervention (no TSSP or MI counselling session).

INTERVENTIONS:
Other: Motivational interviewing counselling session — Individually tailored treatment summary and survivorship care plan provided within a 1-hour 1 hour counseling session with a clinical nurse specialist
  Other Names: MI
  Arms: MI Counselling

SUMMARY:
Treatment summary and survivorship care plans (TSSPs) are poorly studied in Head and Neck Cancer (HNC) patients, and given the high frequency of unmet needs, this patient population has potentially the most to benefit from the implementation of TSSPs. A preliminary feasibility randomized control trial (RCT) at London Regional Cancer Program (LRCP) of 18 patients with HNC evaluating the implementation of TSSPs, found that patients assigned to the intervention group had a 15% higher rate of physician implementation of survivorship care needs compared to the usual care group (40% versus 25%, respectively). Results of the pilot study indicated that successful execution of TSSPs and counselling sessions for HNC patients is feasible. In follow up to the initial feasibility trial, the present investigation seeks to execute a large-scale randomized controlled trial. Three hundred and four patients who were treated at the London Regional Cancer Program (LRCP) for HNC will be randomly assigned to either usual care or a survivorship care plan (TSSP) intervention (90 patients in each arm). The intervention will consist of the delivery of a TSSP and a motivational interviewing counseling session with a clinical nurse specialist tailored to the needs of this vulnerable cancer population. The primary objective of the study is to evaluate the delivery of a TSSP during a one-on-one motivational interviewing counselling session with HNC survivors to determine whether the intervention results in improved implementation of recommendations for HNC survivors compared to usual care. Secondary study objectives will evaluate quality of life and satisfaction with care at 12 months post-intervention between the usual care and intervention group. Primary care providers of patients assigned to the intervention group will also be surveyed on the utility of the TSSP.

DETAILED DESCRIPTION:
This study is a longitudinal randomized controlled trial. Patients will be randomly assigned to either usual treatment or the intervention (MI counselling session). Data will be collected at four time points: baseline (3-6 months post-treatment for HNC), and 3-, 6- and 12- months post-baseline visit. 180 patients with curable stage I-IV head and neck mucosal cancer (HNC) will be recruited to the study (90 per arm).

The intervention will consist of a survivorship care nurse motivational interviewing counseling session coupled with the provision of individualized TSSPs to patients and their health care providers.

The primary outcome will be physician implementation of survivorship care recommendations over the course of 12 months post-intervention assessed by quarterly patient surveys. Secondary outcomes will include adherence to recommended follow-up schedules, quality of life using validated measures, patient satisfaction with care, patient feedback on the utility of the TSSP and counselling session and physician feedback on the utility of the TSSP.

ELIGIBILITY:
Patient Participants

Inclusion Criteria:

* Age 18 years or older
* Willing to provide informed consent
* Diagnosis of stage I-IVA head and neck mucosal cancer (larynx, hypopharynx, oral cavity, oropharynx, nasopharynx)
* Last definitive treatment (surgery, chemotherapy, radiotherapy) between 3 and 6 months prior to enrollment
* English speaking, reading and writing

Exclusion Criteria:

* Second concurrent non-cutaneous malignancy
* Metastatic disease
* Clinically apparent cognitive impairment
* Suspected residual disease after treatment completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Physician implementation of survivorship care recommendations | 12 months
  Physician implementation of survivorship care recommendations over the course of 12 months post-baseline, assessed by quarterly patient reports. Proportion of recommendations implemented by the health care provider will be recorded at 3, 6, and 12-months post-baseline and compared between the intervention and standard care group.

SECONDARY OUTCOMES:
Satisfaction with Care and Information Scale | Baseline, 3, 6, and 12 months post-intervention
  The Satisfaction with Care and Information Scale evaluates participants' level of satisfaction with information provided to them on diagnosis and treatment-related issues, and survivorship issues, using a 5- point Likert scale (1 = very dissatisfied; 5 = very satisfied, range 1 to 5). The means of the responses are calculated to generate satisfaction scores for the following domains: Diagnosis, Oral/dental care, Long-term effects after treatment, Neck/shoulder mobility, Eating/speaking, Post-treatment care, Family/close relationships, and, Overall satisfaction with care and information.
M.D. Anderson Symptom Inventory, Head and Neck Module (MDASI-HN) | Baseline, 3, 6, and 12 months post-intervention
  The MDASI-HN includes a total of 28 items, with sub-scales, including a 13-item core cancer symptoms subscale, a 9-item head and neck-specific symptom subscale, and 6-items assessing the extent that symptoms interfere with daily living. Each item is rated on a 11-point scale from 0 (not at all) to 10 (as bad as you can imagine), while the items that assess the interference of symptoms on daily activities are rated from 0 (does not interfere) to 10 (interfered completely).
Patient Satisfaction with TSSP and Counselling SessionB | Baseline
  Investigator developed survey evaluating patient satisfaction with and feedback on the utility of the TSSP and motivational interviewing counseling session
Physician Satisfaction with TSSP | Baseline
  Investigator developed survey evaluating physician (primary care provider and oncologist) feedback on the utility of the TSSP in addressing head and neck cancer survivorship needs.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle MacNeil, MD, FRCSC, Principal Investigator — Department of Otolaryngology-Head & Neck Surgery, Western University Canada
Locations (1):
- Victoria Hospital, London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Data will be made available upon request

REFERENCES:
- [Derived] Tran B, Dzioba A, Baker J, Mutsaers A, Nichols AC, Mendez A, Goodman CD, Palma DA, Winquist E, Irwin JD, Fung K, Stewart P, Lang P, Correa RJM, Kuruvilla S, Mitchell S, Phillips T, MacNeil SD. The SHARE study - Survivorship After Head and Neck Cancer: evaluating patient care and adherence to follow up in Ontario, Canada: study protocol for a randomized controlled trial. Trials. 2025 Dec 13. doi: 10.1186/s13063-025-09332-5. Online ahead of print. PMID 41390453